CLINICAL TRIAL: NCT05394259
Title: A Pilot Study to Assess the Clinical Utility of PYLARIFY PET-CT for Detecting Metastasis in Pancreatic Cancer, Hepatocellular Carcinoma and Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-1031; NCI-2022-04401 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-05-16; First posted 2022-05-27 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer; Breast Cancer; Hepatocellular Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Breast Neoplasms; Carcinoma, Hepatocellular | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Piflufolastat F18 (Experimental): Piflufolastat F18 will first be given by vein over about 5 seconds.
  Interventions: Drug: Piflufolastat F18

INTERVENTIONS:
Drug: Piflufolastat F18 — Given by vein (IV)
  Other Names: PYLARIFY

SUMMARY:
To learn if piflufolastat F18 can be used in imaging scans for patients with breast cancer, HCC, or pancreatic cancer

DETAILED DESCRIPTION:
Primary Objective:

* To assess the diagnosis accuracy of PYLARIFY (piflufolastat F18 ) PET-CT for imaging patients with suspected metastatic pancreatic cancer, hepatocellular carcinoma (HCC) and breast cancer. Accuracy is defined as the number of concordant cases between PYLARIFY PET-CT and the gold standard truth divided by the total sample size

Secondary Objectives:

* To assess diagnosis accuracy of PYLARIFY (piflufolastat F18 ) PET-CT for imaging patients with suspected metastatic pancreatic cancer, hepatocellular carcinoma (HCC) and breast cancer by additional accuracy measures including sensitivity, specificity, negative predictive value and positive predictive value.
* To evaluate the added clinical usefulness of PYLARIFY (piflufolastat F18) PET-CT for imaging patients with suspected metastatic pancreatic cancer, HCC and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of PYLARIFY in patients <18 years of age, children are excluded from this study.
2. ECOG performance status ≤2 (Karnofsky ≥60%,).
3. Subject or subject's Legally Authorized Representative (LAR) is able to understand, willing and able to provide written informed consent.
4. Patients must have histologically or cytologically confirmed pancreatic ductal adenocarcinoma, HCC and invasive lobular carcinoma
5. Patients with either: a) clinical or radiological (SoC CT, or MRI or FDG PET-CT tests) suspicion of metastatic disease; or b) proven metastatic disease but in whom there is suspicion of an even greater tumor burden that could change therapy approach.
6. Patients with at least one measurable lesion on SoC imaging modality (CT, or MRI, or FDG PET-CT).

   Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.
7. Ability and willingness to undergo biopsy if needed per standard of care for possible metastasis which could change therapy approach. Subject requires further confirmatory diagnostic procedures to confirm PYLARIFY (piflufolastat F18)-PET-CT findings and is planned for: a) Biopsy as SoC; or b) Clinical follow- up as SoC.
8. Either: a) treatment naïve; or b) in active treatment but with suboptimal clinical outcome/response, as determined by treating physicians, and with SoC plan to further biopsy suspected metastatic lesions, PYLARIFY (piflufolastat F18) PET- CT can be performed at least 1 day prior to the planned biopsy.
9. Estimated life expectancy of at least 3 months as determined by the Investigator or treating physician.

Exclusion Criteria:

1. Pregnant or breastfeeding during participation in the study are excluded because: There is no information on the risk of adverse developmental outcomes in pregnant women or animals with the use of piflufolastat F18. All radiopharmaceuticals, including PYLARIFY, have the potential to cause fetal harm depending on the fetal stage of development and the magnitude of the radiation dose; There is no information on the presence of piflufolastat F18 in human milk, the effect on the breastfed infant, or the effect on milk production.
2. History of allergic reactions to PSMA PET radiopharmaceuticals.
3. Patients with psychiatric illness/social situations that would limit compliance with study requirements.
4. Unable to lie flat during or tolerate PET-CT
5. Patients who have had chemotherapy, immunotherapy or radiotherapy within 4 weeks prior to PYLARIFY (piflufolastat F18) injection.
6. Contraindications to PYLARIFY Injection have not been established in humans. None are known or have been observed in nonclinical or clinical studies performed to date. As indicated FDA product labels: Androgen deprivation therapy (ADT) and other therapies targeting the androgen pathway, such as androgen receptor antagonists, may result in changes in uptake of PYLARIFY in prostate cancer. The effect of these therapies on performance of PYLARIFY PET has not been established.
7. Subjects with any medical condition or circumstance that the investigator believes may compromise the safety or compliance of the subject to produce reliable data or completing the study.
8. Patients with other types of pancreatic, hepatic or breast neoplasms will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Accuracy is defined as the number of concordant cases between PYLARIFY PET-CT and the gold standard truth divided by the total sample size. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lu, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org